CLINICAL TRIAL: NCT02062801
Title: Prophylactic Ephedrine to Reduce Fetal Bradycardia After Combined Spinal Epidural Labor Analgesia: a Randomized Double Blind Placebo-controlled Study
Brief Title: Prophylactic Ephedrine and Combined Spinal Epidurals for Labor
Acronym: CEASE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, David Gambling, M.D., Medical Director, Surgical Services, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEASE111199
Record Dates: First submitted 2014-02-07; First posted 2014-02-14 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Labor Pain
Keywords: Combined spinal epidural analgesia, labor, fetal bradycardia
MeSH Terms: conditions — Labor Pain | interventions — Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prophylactic ephedrine (Active Comparator): Ephedrine 10mg iv once at time of combined spinal epidural insertion
  Interventions: Drug: Ephedrine
- Normal saline (placebo) control group (Placebo Comparator): 1ml normal saline intravenously once at time of combined spinal epidural insertion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ephedrine — Patients received additional doses of ephedrine 10mg IV to a maximum of 30mg if BP remained low (<90mmHg systolic) and/was associated with persistent fetal bradycardia or maternal symptoms of dizziness and nausea
  Arms: Prophylactic ephedrine
Drug: Placebo — Patients received normal saline (placebo) administered immediately after combined spinal epidural (CSE) placement
  Arms: Normal saline (placebo) control group

SUMMARY:
The combined spinal epidural (CSE) technique has become increasingly popular for labor pain because of its rapid onset and superior first stage analgesia. However, increased risk for early profound fetal bradycardia (EPFB) following CSE continues to be a concern. Various factors are implicated in the etiology of EPFB but the cause is unknown. Ephedrine administration prior to CSE analgesia may help reduce the risk of EPFB, but to date, nobody has studied the impact of a single dose of intravenous (IV) ephedrine given at the time of CSE administration during labor. The purpose of this study is to measure the incidence of EPFB after combined spinal epidural analgesia using standard definitions. The incidence of EPFB will be compared between patients who receive prophylactic ephedrine or placebo at the time of CSE placement.

DETAILED DESCRIPTION:
Background and explanation of rational:

Epidural analgesia (EA) has been used to provide labor pain relief for over 30 years. The technique has been refined over the past 20 years to provide laboring women with higher quality pain relief, less leg weakness and more control over the administration of the pain relief. Since the early 1990s a combined spinal-epidural (CSE) technique has become more popular because it provides more rapid onset pain relief (1). The Principal Investigator has performed a large randomized blinded study at Sharp Mary Birch Hospital for Women and Newborns to compare the effectiveness of CSE with a standard epidural technique and to describe the incidence of common side effects associated with each of them. These included itching, transient hypotension, motor block and transient fetal heart rate (FHR) abnormalities. It was found that the incidence of profound FHR deceleration was increased in the CSE group: 8.5% vs 4.5% for the standard epidural group, although no poor neonatal outcomes were seen in either group. The question was raised whether prophylactic ephedrine given concomitantly with CSE insertion would reduce the incidence of FHR deceleration, thus reducing a significant side effect associated with this otherwise superior pain relief modality for laboring patients. It is uncertain what causes fetal bradycardia after CSE but it is observed more frequently when high dose intraspinal opioids are used (2). Other potential causes include maternal hypotension associated with rapid onset sympathectomy, uterine tetanic contractions associated with sudden decrease in circulating maternal catecholamines, and rapid decent of the presenting part associated with pelvic floor relaxation. This study is not designed to determine the specific causal mechanism. Ephedrine remains one of the most extensively studied vasopressors used to treat hypotension in the obstetric population (3-5). It has both direct and indirect mechanisms of action, stimulating both alpha- and beta-receptors to increase cardiac output, heart rate and systolic and diastolic blood pressure. In the past both animal and laboratory data have demonstrated that ephedrine preserves uterine artery blood flow and fetal pH to a much better degree than other pressors. However, today it is controversial as to whether neosynephrine is a better option to treat hypotension associated with spinal anesthesia for cesarean delivery (6). Nevertheless, ephedrine has been used for decades for the treatment of maternal hypotension and fetal bradycardia associated with the use of epidural analgesia in laboring women.

Many anesthesiologists use prophylactic ephedrine 10mg intravenously to prevent an anticipated fall in maternal BP. As a consequence the risk of nausea and vomiting associated with hypotension is reduced. It is safe in the absence of maternal heart disease or hypertension.

Ephedrine 10 mg intravenously is used routinely in the labor unit and there is a standing order for the RN to use it to a maximum of 30mg when maternal systolic BP < 90mm Hg. Occasionally, ephedrine 10mg intravenously is used to treat fetal bradycardia in the absence of maternal hypotension.

Kreiser et al. studied 145 deliveries where epidural analgesia was administered (7). The patients were randomly allocated before administration of epidural analgesia to receive an intravenous infusion of 10 mg ephedrine, after epidural induction, followed by a continuous infusion for 60 minutes of 20 mg ephedrine (study group) or to receive no ephedrine (control group). The FHR tracing was evaluated for 20 minutes before and 40 minutes after initiating epidural analgesia. Demographic data and clinical and delivery outcome were assessed and compared between the 2 groups.

They found that Injection of ephedrine significantly reduced the rate of major FHR changes appearing 15-25 minutes after induction of epidural analgesia in the study group compared with the control group (2/72 compared with 11/73, respectively; P = .009). To avoid 1 case of adverse FHR changes, 6.8 women should be treated with ephedrine. Maternal and fetal characteristics and outcome and mode of delivery were similar in the 2 groups. Mean arterial pressure was significantly higher in the study group from the time of analgesia induction and during the subsequent 25 minutes. Maternal heart rate was transiently reduced in the study group only.

Cleary-Goldman et al. evaluated 25mg prophylactic intramuscular (IM) ephedrine vs placebo in a similar setting (8). It was found that IM ephedrine decreased the incidence of maternal hypotension and late fetal heart rate decelerations for one hour after administration, but increased the incidence of fetal tachycardia. However, FHR reactivity was improved.

Clinically, in the center the investigators have not observed that prophylactic ephedrine 10mg intravenously impacts significantly on the fetal heart rate. Although the investigators have used the drug prophylactically for many years, and feel that it is useful in preventing fetal bradycardia, a placebo-controlled trial is needed to prove its advantage in this regard.

Specific objectives:

The investigators propose to study the impact of prophylactic intravenous ephedrine on the incidence of early profound fetal bradycardia following CSE analgesia in healthy parturients.

The investigators plan to conduct a randomized placebo-controlled blinded study comparing the efficacy of 10mg intravenous ephedrine versus an equal volume of normal saline administered immediately after CSE placement.

It was shown in an earlier study at the hospital that the incidence of fetal bradycardia within 30 minutes of a CSE is 8.5%. Profound early fetal bradycardia is defined as a drop in fetal heart rate, within 30 minutes of inducing CSE, to < 90 bpm for > 60 seconds. The investigators predict that ephedrine will reduce the incidence of fetal bradycardia within 30 minutes of a CSE from 8.5% to 4% or less.

Methods:

Trial design This will be a prospective RCT using a placebo control. The numbers of subjects to be studied will be determined after performing a pre-study power analysis. All patients will be term parturients in labor with no health problems or obstetric complications

Participants Inclusion criteria: Ability to speak and understand English; term (37-42 weeks' gestation); cephalic presentation; singleton pregnancy; ASA 3 or less; no pregnancy-induced hypertension; no chronic hypertension; BMI <40; no evidence of pre-epidural fetal heart rate abnormality; no IUGR or low AFI. ASA 1-3 women who request epidural analgesia Informed consent signed upon admission to L&D Exclusion criteria: ASA 4 women, BMI > 39, Contraindication to epidural analgesia, Twin pregnancy, Preterm labor, Severe preeclampsia, Decision to perform CS prior to epidural insertion, Unable to read or speak English, Unable or unwilling to sign the IFC

Interventions This study will occur at Sharp Mary Birch hospital. This will be a triple-blind, prospective, randomized study of healthy women who request labor epidural analgesia. Women will be approached by a nurse or investigator in triage or upon admission to labor and delivery with a description of the study. They will sign an informed consent form prior to randomization into one of the two study groups. An explanation will be given that neither arm of the study is experimental but that both techniques are used routinely at Sharp Mary Birch Hospital at the discretion of the attending anesthesiologist. The only elements of this study that are experimental are the random allocation to one of the two groups and the collection of data for statistical analyses. None of the drugs used are experimental and no tests other than those used in normal clinical practice are required during the study.

Once the woman has signed the IFC she will be randomly assigned to receive either 10mg intravenous ephedrine versus an equal volume of normal saline administered immediately after combined spinal epidural (CSE) placement. CSE will be induced in the sitting position at the L3-4 or L2-3 interspace under strict asepsis. All patients will receive a 500ml intravenous preload of lactated Ringers solution.

CSE: once the epidural space has been located, CSF will be obtained via a 26g GM needle and 3.125mg bupivacaine plus 5mcg fentanyl injected (2.5ml total volume). In both groups, a patient-controlled infusion of epidural bupivacaine 0.125% with 2mcg/ml fentanyl will be started immediately as per usual hospital practice.

Routine hemodynamic monitoring and FHR monitoring will be instituted as per standard hospital protocols. The FHR strips will be analyzed by blinded nurses trained in the interpretation of the strips. They will compare FHR baseline for 10 minutes before CSE and up to 30 minutes after CSE. They will also document instances of EPFB and other FHR abnormalities for up to 30 minutes after CSE. They will use national standard definitions for FHR abnormalities.

Outcomes Data collected will include the incidence of profound early fetal bradycardia as previously defined; lowest and highest BP in first 30 minutes; maximum FHR in first 30 minutes; incidence of tetanic uterine contraction; total dose of ephedrine used during labor; use of nitroglycerin or terbutaline to treat tetanic uterine contraction.

Demographic data collected for research purposes will include: patient age, height, weight, gravidity, parity, gestational age, cervical dilatation at time of epidural request; induced or spontaneous labor, use of oxytocin augmentation, type of delivery (spontaneous vaginal, vacuum, forceps, cesarean) and incidence of emergency cesarean delivery, neonatal weight and Apgar scores at 1 and 5 minutes.

The primary outcome for this study is the effect of prophylactic intravenous ephedrine on the incidence of fetal bradycardia within 30 min of CSE. The secondary outcomes for this study will include: Need for urgent cesarean delivery within 30 min of CSE, incidence of tetanic uterine contraction (tachysystole), and the impact of parity and induction on the incidence of fetal bradycardia after CSE.

Recruitment Patients will be recruited between December 1st 2011 and April 15th 2013

Randomization Randomization will be created by a statistician and upcoming sequences will be concealed from the investigators, particularly those involved with recruitment by the use of sealed opaque envelopes. Randomization will be in groups of 20 and stratified for parity and induction of labor.

Allocation concealment mechanism Sealed opaque envelopes will be used to implement the random allocation sequence Implementation The participants will be enrolled by an L&D nurse or attending anesthesiologist. The random allocation sequence will be generated by a statistician. The participants will be randomly assigned to the next allocation in the sequence.

Blinding Investigator, participant, attending nurse and obstetrician and statistician will all be blinded to allocation. The pharmacist will keep the randomization chart and key.

PHI is a necessary component of this research and will be collected by one of the researchers either at the time of the study or from patient records taken from the clinical computer program or the patients' charts. All data collected will be kept in a private and secure location. Patients will be identified only by their study number and initials

Potential Risks The potential or known risks of combined spinal-epidural analgesia and prophylactic ephedrine administration are explained to all patients prior to induction of analgesia. Alternative means of providing pain relief during labor are described. The risks are outlined in the anesthetic consent form and in a video that the woman watches in her antenatal class or immediately prior to the spinal-epidural induction. The risks include hypotension, itching, transient fetal heart rate changes, leg weakness, post-dural puncture headache, failed epidural, infection at the site of epidural insertion, CNS infection (rare), high epidural block with the potential to cause respiratory compromise (rare), seizures and cardiac arrest from local anesthetic toxicity (rare), temporary mild neurological impairment in the lower limbs and, very rarely, permanent paralysis and death

Risk Management/Confidentiality Adverse effects from either treatment will be managed as per usual clinical practice. The procedures for protecting against the risks to confidentiality and use or disclosure of protected health information, include keeping information stored in a secure location and only identifying subjects by study number and initials.

Potential Benefits There are no specific benefits to be gained by the individual subject, but there may be benefits that accrue to society in general if the study shows a significant advantage to one of the two treatments.

ELIGIBILITY:
Inclusion criteria:

* Ability to speak and understand English
* Term (37-42 weeks' gestation)
* Cephalic presentation
* Singleton pregnancy
* ASA 3 or less
* No pregnancy-induced hypertension
* No chronic hypertension
* BMI <40
* No evidence of pre-epidural fetal heart rate abnormality
* No IUGR or low AFI. ASA 1-3 women who request epidural analgesia Informed consent signed upon admission to L&D

Exclusion Criteria:

* ASA 4 women, BMI > 39
* Contraindication to epidural analgesia
* Twin pregnancy
* Preterm labor
* Severe preeclampsia
* Decision to perform CS prior to epidural insertion
* Unable to read or speak English
* Unable or unwilling to sign the IFC

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 710 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Gambling, MB,BS, Principal Investigator — Anesthesia Services Medical Group
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States

REFERENCES:
- [Background] 1. Gambling DR et al.A randomized study of combined spinal-epidural analgesia versus intravenous meperidine during labor. Anesthesiology 1998; 89: 1336-44. 2. Mardirosoff C et al. Fetal bradycardia due to intrathecal opioids for labour analgesia : a systematic review. BJOG 2002; 109: 274-81. 3.Wright RG et al: The effect of maternal administration of ephedrine on fetal heart rate and variability. Obstet Gynecol.1981; 57: 734-8. 4.Tong C, Eisenach JC: The vascular mechanism of ephedrine's beneficial effect on uterine perfusion during pregnancy. Anesthesiology 1992; 76: 792-8 5.Reidy J, Douglas J: Vasopressors in obstetrics. Anesthesiol Clin. 2008 ;26:75-88, vi- vii. Review. 6. Gambling DR, McLaughlin KR. Ephedrine and phenylephrine use during cesarean delivery. Anesthesiology 2010; 112: 1287-8. 7. Kreiser D et al. The effect of ephedrine on intrapartum fetal heart rate after epidural analgesia. Obstet Gynecol. 2004;104:1277-81. 8. Cleary-Goldman J et al.. Prophylactic ephedrine and combined spinal epidural: maternal blood pressure and fetal heart rate patterns. Obstet Gynecol. 2005; 106: 466-72.
- [Derived] Gambling DR, Bender M, Faron S, Glaser D, Farrell TR. Prophylactic intravenous ephedrine to minimize fetal bradycardia after combined spinal-epidural labour analgesia: a randomized controlled study. Can J Anaesth. 2015 Nov;62(11):1201-8. doi: 10.1007/s12630-015-0450-8. Epub 2015 Aug 14. PMID 26272720

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 710 participants met criteria for eligibility in the study. Of that total, 108 declined to participate in the study, and were excluded prior to random group assignment. This resulted in 602 total participants (301 for each of the intervention groups).
Groups:
- Normal Saline Control Group: 1ml normal saline intravenously once at time of combined spinal epidural insertion
  Placebo
Period: Overall Study
Arm/Group | Prophylactic Ephedrine | Normal Saline Control Group
Started | 301 | 301
Completed | 299 | 297
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylactic Ephedrine | Normal Saline Control Group | Total
Number analyzed (Participants) | 299 | 297 | 596
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6) | 30 (5) | 30 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 299 | 297 | 596
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Early Profound Fetal Bradycardia
Description: Incidence of early profound fetal bradycardia
Time Frame: Within 30 minutes of combined spinal epidural (CSE) placement
Measure: Number; unit: participants
Arm/Group | Prophylactic Ephedrine | Normal Saline Control Group
Number analyzed (Participants) | 299 | 297
participants | 8 | 14
Statistical Analysis 1: Comparison: Prophylactic Ephedrine vs Normal Saline Control Group; Test type: Superiority or Other; p = 0.18, Chi-squared

2. Secondary Outcome: Tetanic (Sustained) Uterine Contraction (TUC)
Description: Incidence of Tetanic (sustained) Uterine Contraction (TUC)
Time Frame: Within 30 minutes of combined spinal epidural (CSE) placement
Measure: Number; unit: participants
Arm/Group | Prophylactic Ephedrine | Normal Saline Control Group
Number analyzed (Participants) | 299 | 297
participants | 58 | 58
Statistical Analysis 1: Comparison: Prophylactic Ephedrine vs Normal Saline Control Group; Test type: Superiority or Other; p = 0.97, Chi-squared

3. Secondary Outcome: Urgent Cesarean Delivery
Description: Incidence of urgent cesarean delivery
Time Frame: Within 30 minutes of combined spinal epidural (CSE) placement
Measure: Number; unit: participants
Arm/Group | Prophylactic Ephedrine | Normal Saline Control Group
Number analyzed (Participants) | 299 | 297
participants | 1 | 2
Statistical Analysis 1: Comparison: Prophylactic Ephedrine vs Normal Saline Control Group; Test type: Superiority or Other; p = .56, Chi-squared

ADVERSE EVENTS:
Arm/Group | Prophylactic Ephedrine | Normal Saline Control Group
Serious Adverse Events (participants affected / at risk) | 0/301 | 0/301
Other Adverse Events (participants affected / at risk) | 0/301 | 0/301

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No